CLINICAL TRIAL: NCT00860548
Title: An Observational, Long-term Follow-up Study of Eligible Individuals Declining To Participate in the Scleroderma Cyclophosphamide or Transplantation (SCOT) Study (SCSSc-02)
Brief Title: SCOT Scleroderma Treatment Alternative Registry (STAR Registry)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT SCSSc-02; SCOT
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Scleroderma, Systemic; Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: currently available therapy in the community — Participants will receive telephone calls every 3 months for approximately 44 months for the purpose of outcome surveys

SUMMARY:
The Scleroderma Cyclophosphamide Or Transplant (SCOT) Trial is a Phase II/III interventional trial comparing two treatments for early, severe scleroderma. These two interventions are high dose immunosuppressive therapy followed by autologous stem cell transplantation and monthly high dose pulse cyclophosphamide (the later for 12 doses). While standard of care might be considered the optimal control arm for a trial such as this one, no such standard of care is available for the population of scleroderma patients defined by the eligibility criteria for this trial. The rheumatologists on the protocol team believe that the SCOT cyclophosphamide regimen represents the best control arm for this study. However, given concerns over use of a treatment arm as a control that has not been established as a standard of care, this registry was established. The registry will be a prospective, observational study of subjects with severe systemic sclerosis (SSc) who are eligible to participate in the Scleroderma Cyclophosphamide or Transplantation (SCOT) Study but are denied insurance coverage or decline to participate prior to randomization. Subjects will be accrued over the same period as the SCOT study. Subjects will follow the course of treatment prescribed by their treating physician with no interference from the registry.

The primary purpose of this study is to document the disease course and outcome in a group of participants who are eligible for the SCOT study, but declined to participate, in order to determine whether their outcome is better, worse, or no different than those who participate in the treatment phase of the trial.

DETAILED DESCRIPTION:
For multiple reasons, the SCOT investigators and the sponsor of the SCOT trial, the Division of Allergy, Immunology, and Transplantation (DAIT) of the National Institute of Allergy and Infectious Diseases (NIAID), determined that it is important to track the course of a 'matched' group of patients, who are not exposed to these treatments but receive currently available therapy in the community. First, such a group will provide information to determine if the SCOT entry criteria do indeed identify these high-risk individuals. More importantly, such a group of patients is likely to be treated with a variety of medical regimens, including some immunosuppressive therapy with cyclophosphamide or other immunosuppressive agents that may modify the natural history of the disease. In evaluating the relative efficacy of the two treatment regimens, it will be important to assess whether outcomes in the subjects treated under the SCOT protocol have outcome profiles that differ from those associated with the matched group of patients treated in the community. One readily available group that meets these criteria are those individuals who are otherwise eligible for the SCOT trial but fail to be randomized because they either decline to participate or are denied insurance coverage to receive the SCOT treatment regimens.

The duration of this trial is 44 months. Participants will be enrolled over the same period as the SCOT trial. Participants will follow the course of treatment prescribed by their treating physician with no interference from the registry. All participant contact, including obtainment of informed consent and telephone interview regarding outcome measurements will be performed by SCOT study personnel at the University of Texas, Houston (one of the SCOT transplant centers). Participants will be contacted by phone every 3 months to determine vital status, record medical and other therapy, and administer the modified Scleroderma Health Assessment Questionnaire (S-HAQ). Medical records will be obtained to verify self-reported medical events.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria

Exclusion Criteria:

* No additional exclusion criteria

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with severe systemic sclerosis who are eligible for the SCOT study, but either decline to participate or are denied insurance coverage, prior to randomization will be invited to participate in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 44 months after subject enrollment
  The events will be defined as any one of the following:
  * Death.
  * Respiratory failure defined as the need for supplementary oxygen; or
  * Renal failure, as defined by chronic dialysis > 6 months or renal transplantation.

SECONDARY OUTCOMES:
Functional status as determined by the Modified Scleroderma Health Assessment Questionnaire (m-HAQ/S-HAQ) | 44 months after subject enrollment
Mortality due to any cause | 44 months after subject enrollment
Medical therapies and procedures (including hospitalizations) | 44 months after subject enrollment
Diagnosis and treatment for pulmonary hypertension | 44 months after subject enrollment
Need for hyperalimentation | 44 months after subject enrollment
Amputation whether surgical or auto-amputation | 44 months after subject enrollment
Hospitalization or surgery | 44 months after subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Mayes, MD, MPH, Study Chair — The University of Texas Health Science Center, Houston; Daniel Furst, MD, Study Chair — UCLA Medical School; Peter McSweeney, MD, Study Chair — Blood and Marrow Transplant Program, Presbyterian/St. Luke's Medical Center, Rocky Mountain Cancer Center; Leslie J. Crofford, MD, Study Chair — University of Michigan; Richard Nash, MD, Study Chair — Fred Hutchinson Cancer Center; Keith Sullivan, MD, Study Chair — Division of Cellular Therapy, Duke University
Locations (1):
- University of Texas, Houston Medical School, Houston, Texas, United States

REFERENCES:
- [Background] Czirjak L, Nagy Z, Szegedi G. Survival analysis of 118 patients with systemic sclerosis. J Intern Med. 1993 Sep;234(3):335-7. doi: 10.1111/j.1365-2796.1993.tb00753.x. PMID 8354987
- [Background] Bulpitt KJ, Clements PJ, Lachenbruch PA, Paulus HE, Peter JB, Agopian MS, Singer JZ, Steen VD, Clegg DO, Ziminski CM, Alarcon GS, Luggen ME, Polisson RP, Willkens RF, Reading JC, Williams HJ, Ward JR. Early undifferentiated connective tissue disease: III. Outcome and prognostic indicators in early scleroderma (systemic sclerosis). Ann Intern Med. 1993 Apr 15;118(8):602-9. doi: 10.7326/0003-4819-118-8-199304150-00005. PMID 8452326
- [Background] Follansbee WP, Zerbe TR, Medsger TA Jr. Cardiac and skeletal muscle disease in systemic sclerosis (scleroderma): a high risk association. Am Heart J. 1993 Jan;125(1):194-203. doi: 10.1016/0002-8703(93)90075-k. PMID 8417518
- [Background] Lee P, Langevitz P, Alderdice CA, Aubrey M, Baer PA, Baron M, Buskila D, Dutz JP, Khostanteen I, Piper S, et al. Mortality in systemic sclerosis (scleroderma). Q J Med. 1992 Feb;82(298):139-48. PMID 1620814
- [Background] Steen VD, Mayes MD, Merkel PA. Assessment of kidney involvement. Clin Exp Rheumatol. 2003;21(3 Suppl 29):S29-31. PMID 12889219
- [Background] Clements PJ, Wong WK, Hurwitz EL, Furst DE, Mayes M, White B, Wigley F, Weisman M, Barr W, Moreland L, Medsger TA Jr, Steen V, Martin R, Collier D, Weinstein A, Lally E, Varga J, Weiner S, Andrews B, Abeles M, Seibold J. Correlates of the disability index of the health assessment questionnaire: a measure of functional impairment in systemic sclerosis. Arthritis Rheum. 1999 Nov;42(11):2372-80. doi: 10.1002/1529-0131(199911)42:113.0.CO;2-J. PMID 10555033
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Scleroderma: Cyclophosphamide Or Transplantation (SCOT) Study — http://www.sclerodermatrial.org/